CLINICAL TRIAL: NCT00929305
Title: Study of the Effect of Low Level Laser Therapy on the Reduction of Chronic Pain Associated With Neck and Shoulder Pain of Musculoskeletal Origin.
Brief Title: Low Level Laser Light Therapy and Chronic Neck and Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ECP-002
Record Dates: First submitted 2009-06-25; First posted 2009-06-29 (Estimated); Results first posted 2013-04-22 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Shoulder Pain; Neck Pain; Musculoskeletal Pain; Musculoskeletal Strain; Musculoskeletal Sprain
Keywords: chronic pain; neck; shoulder; musculoskeletal origin
MeSH Terms: conditions — Shoulder Pain; Neck Pain; Musculoskeletal Pain; Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo laser (Placebo Comparator): inactive laser light
  Interventions: Device: Placebo laser
- Erchonia PL2000 (Active Comparator): The Erchonia PL2000 Laser emits 1 milliWatt (mW) of red (635nm wavelength) light via an electric diode energy source. It is a hand-held device that uses rechargeable batteries or a separate power adapter.
  Interventions: Device: Erchonia PL2000

INTERVENTIONS:
Device: Erchonia PL2000 — The Erchonia PL2000 Laser emits 1 mW of red (635nm wavelength) light via an electric diode energy source. It is a hand-held device that uses rechargeable batteries or a separate power adapter.
  Other Names: Erchonia PL5000; Erchonia EVRL Laser
  Arms: Erchonia PL2000
Device: Placebo laser — Inactive laser light
  Arms: Placebo laser

SUMMARY:
The purpose of this study was to determine whether the application of low level laser light therapy to the neck and shoulder region is effective in reducing chronic neck and shoulder pain of musculoskeletal origin.

DETAILED DESCRIPTION:
Chronic neck and shoulder pain arising from osteoarthritis, chronic muscle spasms or thoracic or cervical spine sprain strain can be seriously debilitating. Currently available treatment options such as pain relief medication, ice pack, massage, physical therapy and chiropractic are typically of limited effectiveness. More permanent options such as surgery are invasive with long recovery periods and side-effects and complications of their own. Low level laser light therapy, with its proven anti-inflammatory ability, offers a simple non-invasive option for the reduction of chronic neck and shoulder pain.

ELIGIBILITY:
Inclusion Criteria:

* Location of pain is on the right and/or left side of the neck and/or shoulder and/or the back of the neck.
* Etiology of pain is osteoarthritis/Degenerative Joint Disorder (DJD); chronic muscle spasms or cervical and thoracic spine sprain strain, determined according to subject medical history, medication use history, previous records review, physical examination of the cervical spine and shoulder.
* Stage of injury is chronic, having prevailed for longer than 30 days.
* Degree of Pain self-rating of 50 or greater on the 0-100 Visual Analog Scale (VAS).
* 18-65 years.

Exclusion Criteria:

* Stage of injury is acute, having prevailed for less than 30 days.
* Known herniated disc injury.
* Any other disease or condition that may cause or contribute to the chronic pain condition.
* Presence of infection or open wound at the treatment areas.
* Use of steroids or narcotics.
* Use of over-the-counter (OTC) medication for the relief of pain within the 24-hour period prior to participating in the treatment phase of the study, or prescription medication for the relief of pain within the 48-hour period prior to participating in the treatment phase of the study.
* pregnant or lactating.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2001-01; Primary Completion 2001-06 (Actual); Study Completion 2001-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory C Roche, DO, Principal Investigator; Douglas D Dedo, MD, Principal Investigator; Edward B Lack, MD, Principal Investigator

REFERENCES:
- See also: FDA 510(k)#K012580 clearance based on the results of this study — http://www.accessdata.fda.gov/cdrh_docs/pdf/K012580.pdf
- See also: FDA 510(k)#K050672 clearance based on this study's results — http://www.accessdata.fda.gov/scripts/cdrh/cfdocs/cfpmn/pmn.cfm?ID=17825

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period was June-July, 2001. Locations were 3 private practice test sites: 2 in California and one in Virginia.
Pre-assignment Details: 14 enrolled participants were subsequently excluded for taking study excluded medications, for having a self-reported pre-treatment pain Visual Analog Score (VAS) of less than 50 and for having a herniated disc injury.
Groups:
- Erchonia PL2000: The Erchonia EVRL Laser emits 1 mw of red (635nm wavelength) light via an electric diode energy source (CDRH Class II). It is a hand-held device that uses rechargeable batteries or a separate AC power adapter.
Period: Overall Study
Arm/Group | Placebo Laser | Erchonia PL2000
Started | 43 | 43
Completed | 43 | 43
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Laser | Erchonia PL2000 | Total
Number analyzed (Participants) | 43 | 43 | 86
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 43 | 43 | 86
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 26 | 49
  Male | 20 | 17 | 37
Location of Pain [Number; unit: participants] — Pain on the right and/or left sides of the neck and/or shoulders, or both.
  participants
    Neck only | 16 | 13 | 29
    Shoulder only | 4 | 7 | 11
    Both Neck & Shoulder | 23 | 23 | 46
Origin of Pain [Number; unit: participants] — Pain originating from one or more of three etiologies: osteoarthritis; muscle spasms, sprain strain.
  participants
    muscle spasms and sprain strain | 26 | 31 | 57
    muscle spasms only | 10 | 5 | 15
    osteoarthritis | 7 | 7 | 14
Baseline Visual Analog Scale (VAS) pain rating [Mean (Standard Deviation); unit: units on a scale] — Participants recorded a self-rating of their degree of pain in the neck-shoulder area before the study treatment was administered on the 0-100 standardized Visual Analog Scale (VAS). The VAS is a 100mm long horizontal line ranging from '0: no pain at all' on one end to '100: worst pain imaginable' on the other end. The participant marked the point along the scale that best represented the level of pain they experienced at that time in the neck-shoulder area. The higher the number marked, the greater the pain level.
  units on a scale | 60.00 (8.60) | 60.21 (9.84) | 60.10 (9.19)
Duration of Pain [Mean (Standard Deviation); unit: months] — Duration in months of chronic pain in the neck and/or shoulder region.
  months | 82.95 (86.14) | 61.74 (77.21) | 72.35 (82.01)

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Whose Self-reported Pain Rating in the Neck and Shoulder Area on the 0-100 Visual Analog Scale (VAS) Decreased by 30% or More From Baseline to One Day After Study Treatment
Description: Participants self-rated the degree of pain experienced in the neck-shoulder region on the 0-100 standardized Visual Analog Scale (VAS) at baseline and one day post-treatment. The VAS is a 100mm long horizontal scale ranging from '0: no pain at all' on one end to '100: worst pain imaginable' on the other end. The participant marked the point along the scale that best showed the pain level they experienced in the neck-shoulder area at each point in time. The higher the number marked, the greater the pain level.
Time Frame: baseline and one day
Measure: Number; unit: participants
Arm/Group | Placebo Laser | Erchonia PL2000
Number analyzed (Participants) | 43 | 43
participants | 5 | 28
Statistical Analysis 1: Comparison: Placebo Laser vs Erchonia PL2000; Test type: Superiority or Other; p < 0.0001, Fisher Exact

2. Secondary Outcome: Range of Motion of the Neck and Shoulders
Time Frame: one day
Reporting Status: Not Posted

3. Secondary Outcome: Muscle Trigger Points of the Cervical Spine
Time Frame: one day
Reporting Status: Not Posted

4. Primary Outcome: Change in Self-reported Pain Rating in the Neck and Shoulder Area on the 0-100 Visual Analog Scale (VAS)From Baseline to One Day Post-treatment
Description: Participants self-rated the degree of pain experienced in the neck-shoulder region on the 0-100 standardized Visual Analog Scale (VAS) at baseline and one day post-treatment. The VAS is a 100mm long horizontal scale ranging from '0: no pain at all' on one end to '100: worst pain imaginable' on the other end. The participant marked the point along the scale that best showed the pain level they experienced in the neck-shoulder area at that point in time. The higher the number marked, the greater the pain level.
Time Frame: baseline and one day
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo Laser | Erchonia PL2000
Number analyzed (Participants) | 43 | 43
units on a scale | -4.34 (14.01) | -28.06 (19.95)
Statistical Analysis 1: Comparison: Placebo Laser vs Erchonia PL2000; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Placebo Laser | Erchonia PL2000
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/43
Other Adverse Events (participants affected / at risk) | 0/43 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No